CLINICAL TRIAL: NCT01897883
Title: Dyslipidemia Management in Chinese Post Stroke Patients
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-NCN-XXX-2013/1
Record Dates: First submitted 2013-07-03; First posted 2013-07-12 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2015-07

CONDITIONS: Brain Ischemia,Stoke
MeSH Terms: conditions — Brain Ischemia

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- One Group: Full Analysis Set (FAS) will be the primary analysis set. All post ischemic stroke patients within 6-12 months from attack (i.e., with inclusion criterion No.2 fulfilled) except the screening failure patients, i.e., those who withdraw from the study once the informed consent is given, will be included in the FAS.

SUMMARY:
The purpose of this study is to provide current and reliable data of dyslipidimia management together with control situation of blood pressure and glucose for post-stroke patients within 6-12 months from attack, and also the association between patient characteristics and control rate of lipids in this population.

It is an non-interventional study, no study specified treatment is required.Approximately 5000 post ischemic stroke patients within 6-12 months from attack will enter into the study. Fifty centres from different regions of China will participate in this study.

DETAILED DESCRIPTION:
This is a multicentre, cross-sectional, observational study, aiming to investigate the prevalence and control situation of dyslipidimia in China post ischemic stroke patients within 6-12 months from attack. Patients will be screened consecutively, eligible subjects will be interviewed by investigator and finish a questionire during the visit. Investigator will collect relevant medical history, physical exam results and lab test results including blood lipid (i.e. Triglyceride, Total Cholesterol, LDL-C, HDL-C) and glucose(HbA1c if available).Approximately 5000 post ischemic stroke patients within 6-12 months from attack will enter into the study. Fifty centres from different regions of China will participate in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female with age ≥ 18 years
2. Post ischemic stroke patients within 6-12 months from attack
3. written informed consent is provided to participant in the study

Exclusion Criteria:

1. Significant medical or psychological condition that make patients can not finish the questionnaire independently or with the aids of his/her legal representatives
2. The patient is or will be in another clinical study
3. Previous enrolment in the present study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Post -ischemic stroke patients within 6-12 months from attack, with age ≥ 18 years old. Subject ( or his legal representative) must demonstrate his or her willingness to participate in the survey and comply with its procedures by signing a written consent. Subjects who are unwilling or unable to provide informed consent will be excluded
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2013-07; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
To observe LDL-C level of China post-stroke patients within 6-12 months from attack | Up to 12 months
  Investigator will collect lab test results including blood lipid (i.e. Triglyceride, Total Cholesterol, LDL-C, HDL-C) during the patient visit.
To observe control rate of LDL-C of China post-stroke patients within 6-12 months from attack | Up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Yong Jun Wang, Principal Investigator — Capital Medical University afffiliated Beijing Tiantan Hospital
Locations (26):
- China (26):
  - Research Site, Beijing, Beijing Municipality
  - Research Site, Guangzhou, Guangdong
  - Research Site, Shenzhen, Guangdong
  - Research Site, Haerbin, Heilongjiang
  - Research Site, Zhengzhou, Henan
  - Research Site, Zhenzhou, Henan
  - Research Site, Wuhan, Hubei
  - Research Site, Changsha, Hunan
  - Research Site, Nanjing, Jiangsu
  - Research Site, Suzhou, Jiangsu
  - Research Site, Changchun, Jilin
  - Research Site, Shenyang, Liaoning
  - Research Site, Jinan, Shandong
  - Research Site, Qingdao, Shandong
  - Research Site, Shanghai, Shanghai Municipality
  - Research Site, Xi’an, Shanxi
  - Research Site, Chengdu, Sichuan
  - Research Site, Chongqing, Sichuan
  - Research Site, Tianjin, Tianjin Municipality
  - Research Site, Hangzhou, Zhejiang
  - Research Site, Ruian, Zhejiang
  - Research Site, Taizhou, Zhejiang
  - Research Site, Wenzhou, Zhejiang
  - Research Site, Beijing
  - Research Site, Guangzhou
  - Research Site, Shanghai

REFERENCES:
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1847&filename=Study_synopsis_updated.pdf